CLINICAL TRIAL: NCT01245530
Title: Probable Alzheimer Type Dementia Compare INM-176 1200~1600mg/Day With Donepezil 5~10mg/Day of Safety and Efficacy to Randomization, Multicenter, Double-blind, Double-dummy, Parallel Phase III Clinical Study
Brief Title: An Efficacy and Safety Study of INM-176 for the Treatment of Patients With Alzheimer Type Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Whanin Pharmaceutical Company (Industry)
Responsible Party: Heesook Nam, Whanin Pharmaceutical Company
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INM-176
Record Dates: First submitted 2010-11-01; First posted 2010-11-22 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Alzheimer Type Dementia
Keywords: Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aricept (Active Comparator): Intervention: Drug: Aricept
  Interventions: Drug: Aricept
- INM-176 (Experimental): Intervention: Drug: INM-176
  Interventions: Drug: INM-176

INTERVENTIONS:
Drug: Aricept — Aricept Comparator Intervention: Drug: Aricept 5~10 mg orally every day for 24weeks
  Other Names: Donepezil HCl
  Arms: Aricept
Drug: INM-176 — INM-176: Experimental Intervention: Drug:INM-176 600~1200 mg orally every day for 24weeks
  Other Names: KR-WAP-026
  Arms: INM-176

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two fixed dose (1200mg/day, 1600mg/day) of INM-176 (a drug of treating dementia) comparing with donepezil for treatment for patients with Alzheimer type dementia.

DETAILED DESCRIPTION:
Probable Alzheimer type dementia compare INM-176 1200~1600mg/day with Donepezil 5~10mg/day of safety and efficacy to randomization, multicenter, double-blind, double-dummy, parallel Phase III clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age range : 50 ~ 80 years old
2. Informed consent signed and dated by patient or legal representative
3. Subjects diagnosed with Alzheimer's disease according to DSM-IV criteria
4. Subjects diagnosed with probable Alzheimer's disease according to the National Institute of Neurological and Communicative Disorders and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
5. MMSE score 10 to 26
6. CDR(Clinical Dementia Rating) score 1~2 or GDS(Global Deterioration Scale) 3~5 stage
7. Subjects who didn't take any medication for AchEI (donepezil, memantine, galantamin, etc) before treating or can stop medication at least 4 weeks more prior to screening visit
8. Subjects menopause women or her/his spouse consent with contraception during the study period and 90 days after end of study

Exclusion Criteria:

1. Subjects with psychiatric disorders other than Alzheimer's disease, such as schizophrenia, depression, bipolar disorder, etc
2. Subjects diagnosed or accompanied with Dementia due to other Neurodegenerative disorders (AIDS, syphilis, creutzfeldt-jacob disease, Picks Disease, Huntingtons Disease, Parkinsons disease related dementia)
3. Subjects diagnosed with vascular dementia
4. Subjects diagnosed with stroke within last 3 months prior to screening visit
5. Subjects who have medical history of significant hepatic disease in screening visit (2 ULN≤ALT, AST)
6. Subjects who have medical history of significant renal disease in screening visit (1.5mg/dl≤Serum creatinine)
7. Subjects who have difficult with regulating blood glucose level with anti-diabetes drug (8.0%<HbA1c)
8. Subjects who have medical history of myocardial infarction or arrhythmia
9. Subjects who take warfarin with Atrial fibrillation
10. Pregnant or nursing women
11. Subjects who p0articipated in other clinical trail within last 3 months
12. Subjects who have hypersensitivity to AchEl (acetylcholinesterase inhibitor)
13. Subjects who have unstable clinical laboratory result in screening visit
14. Subjects doubted the pulmonary disease on the chest X-ray in screening visit
15. Subjects considered unsuitable to participate in clinical trail by investigator

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2008-06; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in cognition as assessed by the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) total score | up to 24 weeks

SECONDARY OUTCOMES:
Change from baseline to endpoint in Mini-Mental State Examination (MMSE) | up to 24 weeks
Change from baseline to endpoint in Clinical Dementia Rating | up to 24 weeks
Change from baseline to endpoint in Global Deterioration Scale(GDS) | up to 24 weeks
Change from baseline to endpoint in Korean Activity of Living(K-IADL) | up to 24 weeks
Change from baseline to endpoint in Korean Neuropsychiatric Inventory (NPI) | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SangYoon Kim, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Whanin Pharm.Co.,Ltd., Seoul, Moonjung, South Korea